CLINICAL TRIAL: NCT03301012
Title: Smartphone Addiction Recovery Coach for Young Adults (SARC-YA) Experiment
Acronym: SARC-YA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chestnut Health Systems (Other)
Responsible Party: Principal Investigator, Michael L. Dennis, Ph.D., Senior Research Psychologist and GAIN Coordinating Center Director, Chestnut Health Systems
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DA011323-15
Record Dates: First submitted 2017-09-27; First posted 2017-10-04 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Substance Use Disorders
Keywords: Young Adults; Relapse Prevention; Smartphone; Recovery Support
MeSH Terms: conditions — Substance-Related Disorders | interventions — Secondary Prevention

STUDY DESIGN:
Intervention Model Description: Participants in the control and experimental condition will have access to post treatment recovery support services as usual.
  Participants in the experimental condition will receive a smartphone, a calling/texting/data plan, and the SARC-A mobile applications for the first 6 months post treatment discharge. Experimental participants will 1) complete a 2-3 minute recovery-focused ecological momentary assessment (EMA) at 5 random times a day, receive feedback on their current answers, and provided access to behavioral charting of their past answers over time; and 2) receive continuous access to a suite of self-initiated ecological momentary interventions (EMI) to support their recovery via tool box of coping tools, apps related to getting support, and apps related to maintaining a healthy lifestyle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery Support as Usual Control (Active Comparator): Participants in the control and experimental condition will have access to post treatment recovery support services as usual.
  Interventions: Other: Recovery support as usual; Other: Smartphone assisted relapse prevention
- Smartphone Addiction Recovery Coach (SARC) - Assisted Relapse Prevention (Experimental): Participants in the experimental condition will receive a smartphone, a calling/texting/data plan, and the SARC-YA mobile applications for the first 6 months post treatment discharge. Experimental participants will 1) complete a 2-3 minute recovery-focused ecological momentary assessment (EMA) at 5 random times a day, receive feedback on their current answers, and provided access to behavioral charting of their past answers over time; and 2) receive continuous access to a suite of self-initiated ecological momentary interventions (EMI) to support their recovery via tool box of coping tools, apps related to getting support, and apps related to maintaining a healthy lifestyle.
  Interventions: Other: Smartphone assisted relapse prevention

INTERVENTIONS:
Other: Recovery support as usual — same as arm
  Arms: Recovery Support as Usual Control
Other: Smartphone assisted relapse prevention — same as arm
  Other Names: Relapse Prevention

SUMMARY:
At discharge from outpatient treatment, researchers will recruit 300 young adults and randomly assign them to recovery support as usual control condition or the Smartphone Addiction Recovery Coach for Young Adults (SARC-YA) experimental condition. Participants in the experimental conditions will receive a smartphone, a calling/texting/data plan, and the SARC-YA mobile applications for the first 6 months post treatment discharge. Experimental participants will 1) complete a 2-3 minute recovery-focused ecological momentary assessment (EMA) at 5 random times a day, receive feedback on their current answers, and provided access to behavioral charting of their past answers over time; and 2) receive continuous access to a suite of self-initiated ecological momentary interventions (EMI) to support their recovery via tool box of coping tools, apps related to getting support, and apps related to maintaining a healthy lifestyle. Data include standardized assessments, urine tests, mobile phone metadata, EMA responses, and EMI utilization. The study's primary aim and hypothesis are:

Aim 1: Test the effects of experimental assignment on the frequency of substance use.

H1 Relative to the control group, participants in the experimental group will have lower scores on the quarterly Substance Frequency Scale (3, 6, 9 months post- discharge).

DETAILED DESCRIPTION:
At discharge from outpatient treatment, researchers will recruit 300 young adults and randomly assign them to recovery support as usual control condition or the Smartphone Addiction Recovery Coach for Young Adults (SARC-YA) experimental condition. Participants in the experimental conditions will receive a smartphone, a calling/texting/data plan, and the SARC-YA mobile applications for the first 6 months post treatment discharge. Experimental participants will 1) complete a 2-3 minute recovery-focused ecological momentary assessment (EMA) at 5 random times a day, receive feedback on their current answers, and provided access to behavioral charting of their past answers over time; and 2) receive continuous access to a suite of self-initiated ecological momentary interventions (EMI) to support their recovery via tool box of coping tools, apps related to getting support, and apps related to maintaining a healthy lifestyle. Data include standardized assessments, urine tests, mobile phone metadata, EMA responses, and EMI utilization. The study's aims and their associated hypotheses are:

Aim 1: Test the effects of experimental assignment on the frequency of substance use.

H1 Relative to the control group, participants in the experimental group will have lower scores on the quarterly Substance Frequency Scale (3, 6, 9 months post- discharge). Aim 2: Evaluate the extent to which the experimental effects are moderated by baseline substance use frequency. H2 The Substance Frequency Scale Scores at intake will moderate the effects of experimental on the quarterly subsequent Substance Frequency Scale scores. Aim 3: Test the extent to which the frequency of substance use mediates the effects of experimental assignment on other aspects of recovery including SUD symptoms, HIV risk behavior, quality of life, mental wellness, and days of school. H3a Relative to the control group, participants in the experimental group will have better scores on other aspects of recovery (reverse of number of SUD symptoms, reverse of HIV risk behaviors, quality of life, mental wellness, days of school) in the quarterly interviews. H3b Higher Substance Frequency Scale scores (regardless of assignment) in a given quarter will be associated with worse scores on other aspects of recovery in the next quarter. H3c Substance Frequency Scale scores in a given quarter will mediate the impact of the experimental assignment on other aspects of recovery in the next quarter. Aim 4: Within the experimental condition, determine the degree to which EMA responses (e.g., use, withdrawal, craving, negative and positive affect) and EMI utilization predict the duration of abstinence (to be done within experimental condition.) H4a The duration of abstinence will be negatively related to EMA measures of the recency of use, withdrawal, craving, low self-efficacy to resist relapse, increased negative affect, and decreased positive affect. H4b The duration of abstinence will be positively related to immediate and cumulative EMI utilization.

ELIGIBILITY:
Inclusion Criteria:

1. discharge from an adolescent outpatient SUD treatment program to the community;
2. substance use during the 90 days prior to treatment;
3. aged 18 to 26 at the time of discharge;

   Exclusion Criteria:
4. inability to read and communicate in English;
5. does NOT reside or plan to stay in Chicago during the next 9 months;

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 237 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in GAIN's Substance Frequency Scale from baseline to 6 months (effect of providing the intervention) | 6 month SFS minus baseline SFS
  The GAIN's Substance Frequency Scale (SFS; alpha=.85; test-retest rho=.94) ranges from 0 to 100% and is calculated as the average percent of days in the past 90 that adolescents reported alcohol, cannabis, stimulates, opioids, and other substance use, days of heavy substance use, and days of problems from substance use. Thus it incorporates the frequency of use, range of substances used, amount used, and degree to which use is causing problems.

SECONDARY OUTCOMES:
Change in GAIN's Substance Frequency Scale from 6 to 9 months (effect of withdrawing the intervention) | 9 months SFS minus 6 month SFS
  The GAIN's Substance Frequency Scale (SFS; alpha=.85; test-retest rho=.94) ranges from 0 to 100% and is calculated as the average percent of days in the past 90 that adolescents reported alcohol, cannabis, stimulates, opioids, and other substance use, days of heavy substance use, and days of problems from substance use. Thus it incorporates the frequency of use, range of substances used, amount used, and degree to which use is causing problems.
Change in GAIN Substance Disorder Screener (SDScr) from baseline to 6 months | 6 month minus baseline
  Count of 5 past 90 day substance use disorder symptoms (alpha=.90) from the GAIN-Q3
Change in GAIN Risk Behavior Screener (RBScr) from baseline to 6 months | 6 month minus baseline
  Count of 6 past 90 day of HIV risk behaviors (test-retest rho=.80) including needle use, needle sharing, unprotected sex, multiple sexual partners, trading sex, and victimization from the GAIN-Q3
Change in European Quality of Life 5 dimensions (EQ5D) from baseline to 6 months | 6 month minus baseline
  Count of 6 quality of life items (alpha=.83) from the EQ5D
Change in Mental Health Continuum Short Form (MHC-SF) from baseline to 6 months | 6 month minus baseline
  Count of 14 items related to mental wellness (alpha=.94) from the MHC-SF
Change in the days of school from baseline to 6 months | 6 month minus baseline
  The days of being in school during the past quarter (test-retest rho=.88) from the GAIN-Q3
Duration of abstinence after a given EMA | Measured at 5 random times per day over 6 months in the experimental condition
  The duration of abstinence is the time from each completed EMA to the next indication of use - measured in days.

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Dennis, Ph.D., Principal Investigator — Chestnut Health Systems
Locations (2):
- United States (2):
  - Chestnut Health Systems, Bloomington, Illinois
  - Chestnut Health Systems, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided
We use standardized measures and have a history of established relationships with several investigators who have had their own funds to conduct secondary analyses or need very limited support and are open to others. For EMA/EMI data from the pilot (and for this study, if funded) we are explicitly collaborating with Dr. Susan Murphy at the University of Michigan in her efforts to develop and evaluate Machine Learning algorithms on how to increase EMI utilization and prevent relapse even more effectively. Our data sharing practices have and will continue to include a mixture of publishing traditional peer-reviewed publications; making forms, reports, and normative tables available via the internet (or by request); providing analytic runs upon request; collaborating with other researchers; and providing copies of the de-identified data sets to eligible researchers. The later require data sharing agreements and commitments not to attempt re-identification.

DOCUMENTS (1):
  • Informed Consent Form (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT03301012/ICF_000.pdf